CLINICAL TRIAL: NCT05552261
Title: A Long-term Extension Study to Evaluate the Safety and Efficacy of OXERVATE® 0.002% (20 mcg/mL) Cenegermin-bkbj Ophthalmic Solution in Patients With Stage 1 Neurotrophic Keratitis Who Enrolled in the DEFENDO Study (NGF0120)
Brief Title: DEFENDO Long Term Follow-up Study in Stage 1 NK Patients
Status: Completed | Type: Observational
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Other Study IDs: NGF0122
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Neurotrophic Keratitis
Keywords: Stage 1 NK; OXERVATE®; Cenegermin; NK; DEFENDO; NGF0120 (original DEFENDO study); NGF0122 (DEFENDO long-term follow-up study)
MeSH Terms: interventions — cenegermin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group Long-term follow-up: All eligible patients, after completing enrollment in the original DEFENDO Study, were invited to enter the DEFENDO Long-Term Follow-Up Study (all standard of care permitted), according to inclusion and exclusion criteria.
  Interventions: Drug: Cenegemin in the DEFENDO Study

INTERVENTIONS:
Drug: Cenegemin in the DEFENDO Study — Cenegemin as administered in the original DEFENDO Study. Long-term safety and efficacy of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution administered in Stage 1 Neurotrophic Keratitis (NK) patients enrolled in the original DEFENDO Study (NGF0120 / NCT04485546).
  No intervention was performed in this follow-up / extension study.
  Other Names: OXERVATE®

SUMMARY:
Primary Objective

To evaluate the long-term safety and efficacy (healing) of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution in Stage 1 neurotrophic keratitis (NK) patients who enrolled in the DEFENDO study.

Secondary Objective

To evaluate the long-term efficacy of OXERVATE® 0.002% (20 mcg/mL) cenergemin-bkbj ophthalmic solution in terms of corneal sensitivity, Schirmer I test, tear film break-up time (TFBUT), best corrected distance visual acuity (BCDVA), and quality of life at 24 and 30 months post-treatment

DETAILED DESCRIPTION:
NGF0122 (DEFENDO Long-Term Follow-up) study was a Phase 4, multicenter, open label, long-term follow-up study evaluating safety and efficacy in the patients with Stage 1 Neurotrophic Keratitis (NK) who were enrolled in the NGF0120 (original DEFENDO) study and were treated with OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophthalmic solution for up to 8 weeks in the NGF0120.

After completing enrollment in the NGF0120 Study, patients were invited to enter the NGF0122 Study (all standard of care permitted) in which two additional long-term follow-up visits occurred at 24- and 30-months post-treatment to evaluate long-term clinical outcomes.

In the NGF0122, study patients enrolled in the NFG0120 study were evaluated starting from week 8, which corresponds to the end of treatment of the NGF0120 study and is to be considered as the baseline of the NGF0122 study itself.

Patients were treated per standard of care including additional OXERVATE® 0.002% if deemed appropriate by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Previously enrolled in the DEFENDO Study.
2. Satisfied all Informed Consent requirements. The patient and/or their legal representative read, signed, and dated the IRB approved Informed Consent document before any study-related procedures were performed.
3. Had the ability and willingness to comply with study procedures.

Exclusion Criteria:

Were participating in another study that involved treating the study eye. Participation in non-ocular studies was acceptable provided that the treatment was not considered to be confounding with the DEFENDO Long-Term Follow-up Study, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 1 NK
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD, PhD, Study Chair — Dompé
Locations (4):
- United States (4):
  - New Vision Institute, San Diego, California
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Scheie Eye Institute, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 37 patients enrolled in the original NGF0120 (DEFENDO) study, 24 patients chose to enroll in the long-term follow-up study (henceforth, "extension study", or "long-term follow-up study", NGF0122). All 24 patients had data available at the Month 24 visit, at the Month 30 visit, or both and were included in the FAS.
Groups:
- Group Long-term Follow-up: All eligible patients in the original NGF0120 study, after completing enrollment, were invited to enter the Long- Term Follow-up Study (NGF0122)(all standard of care permitted), according to inclusion and exclusion criteria.
  The NGF0122 study aim was to assess the safety and efficacy of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophtalmic solution administered in Stage 1 Neurotrophic Keratitis patients enrolled in the original NGF0120 study. No intervention was performed in this extension study.
Period: Overall Study
Arm/Group | Group Long-term Follow-up
Started | 24
FAS Set (The FAS (N=24) was the only analysis population in the extension study used for both efficacy and safety analyses. The FAS included all enrolled patients who attended either the Month 24 or Month 30 study visit or both in this extension study.) | 24
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Failure to return to the study clinic within the allowed study window for the Month 30 visit | 2

BASELINE CHARACTERISTICS:
Population: FAS population: The FAS (N=24) was the only analysis population in the extension study used for both efficacy and safety analyses. The FAS included all enrolled patients who attended either the Month 24 or Month 30 study visit or both in this extension study.
Groups:
- Group Long-term Follow-up - FAS: All eligible patients in the original NGF0120 study, after completing enrollment, were invited to enter the Long-Term Follow-up Study (NGF0122)(all standard of care permitted), according to inclusion and exclusion criteria.
  The NGF0122 study aim was to assess the safety and efficacy of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophtalmic solution administered in Stage 1 Neurotrophic Keratitis patients enrolled in the original NGF0120 study.
  No intervention was performed in this extension study.
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Number/Percentage of Patients Who Achieved Corneal Epithelial Healing at NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) and Remained Healed at Month 24 and Month 30 of the NGF0122 Study
Description: Corneal epithelial at Month 24 and Month 30 of the NGF0122 study was summarized as a binary goal attainment variable (Yes/No) based on the subset of patients who achieved corneal epithelial healing at Week 8 of the NGF0120, as determined by the Central Reading Center (CRC).
  Healing was defined as the absence of persistent epithelial staining abnormalities related to disease.
  The persistence (or worsening) of a staining pattern in the same corneal area was considered a failure in terms of healing.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: The Full Analysis Set (FAS) included all enrolled patients who attended either the Month 24 or Month 30 study visit or both in this extension study. The FAS was used for both efficacy and safety analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
Participants
  Healed at NGF0120 Week 8 | 22
  Remained healed at month 24: number analyzed (Participants) | 17
  Remained healed at month 24 | 14
  Remained healed at month 30: number analyzed (Participants) | 20
  Remained healed at month 30 | 16

2. Primary Outcome: Number/Percentage of Patients Who Did Not Achieve Corneal Epithelial Healing at NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) Who Had a Healed Corneal Epithelium at Month 24 and 30 of the NGF0122 Study.
Description: Corneal epithelial healing at the overall Follow-up Month 24 and Month 30 was summarized as a binary goal attainment variable (Yes/No) based on the subset of patients who did not achieve corneal epithelial healing at Week 8 of the NGF0120, as determined by the Central Reading Center (CRC). Healing was defined as the absence of persistent epithelial staining abnormalities related to disease.
  Epithelial healing took into consideration the Baseline epithelial staining patterns of each patient and their evolution over time.The persistence (or worsening) of a staining pattern in the same corneal area was considered a failure in terms of healing.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: The Full Analysis Set (FAS) included all enrolled patients who attended either the Month 24 or Month 30 study visit or both in this extension study. The FAS was used for both efficacy and safety analyses.
  Please note that while at the Month 24 visit both patients had available data, at the month 30 only one of the two patients had available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
Participants
  Not healed at NGF0120 Week 8 | 2
  Healed at month 24: number analyzed (Participants) | 2
  Healed at month 24 | 2
  Healed at month 30: number analyzed (Participants) | 1
  Healed at month 30 | 1

3. Secondary Outcome: Number/Percentage of Patients With an Improvement in Corneal Sensitivity at NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) Who Still Had Improvement in Corneal Sensitivity at Month 24 and 30 of the NGF0122 Study.
Description: Improvement in corneal sensitivity at the overall Follow-up Month 24 and 30 was assessed as a binary goal attainment variable (Yes/No), based on the subset of patients who achieved an improvement in corneal sensitivity at Week 8 of the NGF0120. Improvement was defined as a change from Baseline > 0 cm in the study eye. Corneal sensitivity was measured in the central National Eye Institute (NEI) zone using the Cochet-Bonnet aesthesiometer, before the instillation of any dilating or anesthetic drops. The filament was extended to its full length (6 cm), then retracted in 0.5 cm increments until the patient reported feeling contact. The filament length at which sensation was reported was recorded. Higher values indicate better sensitivity. Please note that patients without a Yes/No response available (=missing data) are not considered in the analysis. More in details, these missing patients are 4 at month 24 and 3 at month 30.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
Participants
  Number of patients improved at Week 8 of the NGF0120 study | 22
  Still had improvement at month 24: number analyzed (Participants) | 18
  Still had improvement at month 24 | 11
  Still had improvement at month 30: number analyzed (Participants) | 20
  Still had improvement at month 30 | 14

4. Secondary Outcome: Number/Percentage of Patients Who Did Not Improved Corneal Sensitivity at NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) and Improved Corneal Sensitivity at Month 24 and 30 of the NGF0122 Study.
Description: Improvement in corneal sensitivity at the overall Follow-up Month 24 and 30 was assessed as a binary goal attainment variable (Yes/No), based on the subset of patients who did not achieve an improvement in corneal sensitivity at Week 8 of the NGF0120. Improvement was defined as a change from Baseline > 0 cm in the study eye. Corneal sensitivity was measured using the Cochet-Bonnet aesthesiometer in the central NEI zone before the instillation of any anesthetic or dilating drops. The filament was extended to 6 cm and retracted in 0.5 cm increments until the patient reported sensation upon contact. Higher values indicate better sensitivity. Please note that patients without a Yes/No response available (=missing data) are not considered in the analysis. More in details, these missing patients are 1 at month 30 only.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
Participants
  Number of patients not improved at Week 8 of the NGF0120 | 2
  Had improvement at month 24: number analyzed (Participants) | 2
  Had improvement at month 24 | 1
  Had improvement at month 30: number analyzed (Participants) | 1
  Had improvement at month 30 | 0

5. Secondary Outcome: Mean Change in Corneal Sensitivity From NGF0120 Baseline and NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) to Month 24 and Month 30 of the NGF0122 Study.
Description: Corneal sensitivity at the overall Follow-up Month 24 and Month 30 measured (in cm) in the qualifying NEI (National Eye Institute) zone of the study eye using the Cochet-Bonnet aesthesiometer before the instillation of any anesthetic or dilating drops.
  Improvement was defined as a change from Baseline > 0 cm in the study eye. Higher values indicate better sensitivity.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
cm
  Change from Baseline to month 24: number analyzed (Participants) | 20
  Change from Baseline to month 24 | 1.03 (1.853)
  Change from week 8 to month 24: number analyzed (Participants) | 20
  Change from week 8 to month 24 | -0.69 (1.953)
  Change from Baseline to month 30: number analyzed (Participants) | 21
  Change from Baseline to month 30 | 1.21 (1.743)
  Change from week 8 to month 30: number analyzed (Participants) | 21
  Change from week 8 to month 30 | -0.63 (1.816)

6. Secondary Outcome: Change From NGF0120 Baseline and NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) in Schirmer I Scores to Month 24 and Month 30 of the NGF0122 Study.
Description: Change in Schirmer I test scores was assessed as a continuous outcome in the study eye from Baseline and at Week 8 of the NGF0120 to Month 24 and Month 30.
  The Schirmer I test was conducted on unanesthetized eyes using standardized paper test strips placed in the lower temporal lid margin of each eye. After 5 minutes, the strip was removed, and the length of the moistened area (in millimeters) was recorded.This test measures aqueous tear production. Any change in mean score >0 was considered an improvement in dry eye. Higher scores indicate better tear production, while lower values are associated with more severe dry eye. A positive change from Baseline was interpreted as improvement.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
mm
  from baseline to month 24: number analyzed (Participants) | 20
  from baseline to month 24 | -2.8 (8.55)
  from week 8 to month 24: number analyzed (Participants) | 20
  from week 8 to month 24 | -4.9 (9.13)
  from baseline to month 30: number analyzed (Participants) | 20
  from baseline to month 30 | -0.8 (7.69)
  from week 8 to month 30: number analyzed (Participants) | 20
  from week 8 to month 30 | -3.1 (5.35)
Statistical Analysis 1: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.5158, Wilcoxon signed-rank; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-6.7 to 1.2]
Statistical Analysis 2: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.0670, Wilcoxon signed-rank; Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-9.2 to -0.6]
Statistical Analysis 3: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.6307, Wilcoxon signed-rank; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-4.4 to 2.8]
Statistical Analysis 4: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.0357, Wilcoxon signed-rank; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-5.6 to -0.6]

7. Secondary Outcome: Change From NGF0120 Baseline and NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) in TFBUT to Months 24 and 30 of the NGF0122.
Description: Change in Tear Film Break-Up Time was evaluated in the study eye. TFBUT was measured in seconds using fluorescein dye under cobalt blue illumination. After fluorescein instillation, the patient blinked once or twice, then kept the eye open; the time to first dry spot was recorded. Two values were averaged, or three if differing by >2 seconds. TFBUT values ranged from 0 seconds (tear film instability) to ≥10 seconds (normal stability). Values <5 seconds suggest clinically relevant tear film dysfunction. A positive change from Baseline or Week 8 (>0 seconds) was interpreted as improvement in tear film stability.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
sec
  From baseline to month 24: number analyzed (Participants) | 20
  From baseline to month 24 | 0.695 (2.2390)
  From week 8 to month 24: number analyzed (Participants) | 20
  From week 8 to month 24 | 0.539 (2.3275)
  From baseline to month 30: number analyzed (Participants) | 21
  From baseline to month 30 | -0.384 (2.0018)
  From week 8 to month 30: number analyzed (Participants) | 21
  From week 8 to month 30 | -0.561 (2.2242)
Statistical Analysis 1: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.2836, Wilcoxon signed-rank; Mean Difference (Final Values) = 0.695, 95% CI 2-sided [-0.353 to 1.743]
Statistical Analysis 2: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.5153, Wilcoxon signed-rank; Mean Difference (Final Values) = 0.539, 95% CI 2-sided [-0.550 to 1.628]
Statistical Analysis 3: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.2530, Wilcoxon signed-rank; Mean Difference (Final Values) = -0.384, 95% CI 2-sided [-1.295 to 0.527]
Statistical Analysis 4: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.3828, Wilcoxon signed-rank; Mean Difference (Final Values) = -0.561, 95% CI 2-sided [-1.574 to 0.451]

8. Secondary Outcome: Number/Percentage of Patients Who Achieved a 15-letter Improvement in BCDVA From NGF0120 Baseline and NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) to Month 24 and Month 30 of the NGF0122 Study.
Description: Best Corrected Distance Visual Acuity (BCDVA) at the overall Follow-up Month 24 and Month 30 was assessed in the study eye using the ETDRS visual acuity chart at a distance of 4 meters (13.1 feet), prior to any administration of anesthetic or mydriatic eye drops. Results were recorded as the number of letters correctly identified on the chart. This outcome evaluated the number and percentage of patients who gained at least 15 letters in BCDVA from DEFENDO Baseline and week 8, at Month 24 and Month 30. A gain of ≥15 letters is considered a clinically meaningful improvement corresponding to approximately three lines on the ETDRS chart. The endpoint was analyzed as a binary variable (Yes/No).
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
Participants
  Achieved a 15-letter Gain from Baseline to month 24: number analyzed (Participants) | 20
  Achieved a 15-letter Gain from Baseline to month 24 | 2
  Achieved a 15-letter Gain from Baseline to month 30: number analyzed (Participants) | 21
  Achieved a 15-letter Gain from Baseline to month 30 | 1
  Achieved a 15-letter Gain from Week 8 to month 24: number analyzed (Participants) | 19
  Achieved a 15-letter Gain from Week 8 to month 24 | 0
  Achieved a 15-letter Gain from Week 8 to month 30: number analyzed (Participants) | 20
  Achieved a 15-letter Gain from Week 8 to month 30 | 0

9. Secondary Outcome: Change From NGF0120 Baseline and NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) to Month 24 and Month 30 of the NGF0122 Study.
Description: Best Corrected Distance Visual Acuity (BCDVA) at Month 24 and Month 30 was assessed in the study eye using the ETDRS visual acuity chart at 4 meters (13.1 feet), before any anesthetic or mydriatic eye drops or ocular procedures. Scores were recorded in logMAR units, ranging from -0.3 (better visual acuity) to 1.0 (poorer acuity). Higher logMAR values indicate worse vision. A negative change in logMAR (i.e., <0) indicated an improvement in visual acuity. Mean values and standard deviations were summarized descriptively at each timepoint.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
score on a scale
  From baseline to month 24: number analyzed (Participants) | 20
  From baseline to month 24 | -0.023 (0.1855)
  From week 8 to month 24: number analyzed (Participants) | 19
  From week 8 to month 24 | 0.124 (0.1097)
  From baseline to month 30: number analyzed (Participants) | 21
  From baseline to month 30 | -0.056 (0.1705)
  From week 8 to month 30: number analyzed (Participants) | 20
  From week 8 to month 30 | 0.087 (0.1440)
Statistical Analysis 1: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.7450, Wilcoxon signed-rank; Mean Difference (Final Values) = -0.023, 95% CI 2-sided [-0.110 to 0.064]
Statistical Analysis 2: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p < 0.0001, Wilcoxon signed-rank; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.071 to 0.177]
Statistical Analysis 3: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.1619, Wilcoxon signed-rank; Mean Difference (Final Values) = -0.056, 95% CI 2-sided [-0.134 to 0.021]
Statistical Analysis 4: Comparison: Group Long-term Follow-up - FAS; Test type: Other; p = 0.0100, Wilcoxon signed-rank; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [0.020 to 0.154]

10. Secondary Outcome: Change From NGF0120 Baseline and NGF0120 Week 8 (EoT NGF0120 = Baseline NGF0122) in Quality of Life (QoL) Expressed by the IDEEL to Months 24 and 30 of the NGF0122 Study.
Description: "Impact of Dry Eye on Everyday Life" (IDEEL) is a 57-item questionnaire assessing dry eye impact (and consequently QoL), composed by 6 domains:
  * Daily Activities; Higher score = less impact
  * Emotional Impact: Higher score = less impact on emotions
  * Impact on Work: Higher score = less impact on work
  * Symptom Bother: Higher score = greater symptom bother
  * Treatment Bother: Higher score = less treatment-related bother
  * Treatment Effectiveness: Higher score = greater satisfaction with treatment effectiveness For 5 of 6 domains (Symptom Bother), higher scores on a 0-100 scale indicated improved quality of life relative to dry eye symptoms. For the domain of "symptom bother", a higher score indicated greater symptom bother. For this reason no total score, but only subscores, is calculated.
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
score on a scale
  Daily activities - from baseline to month 24: number analyzed (Participants) | 21
  Daily activities - from baseline to month 24 | -0.32 (18.466)
  Daily activities - change from week 8 to month 24: number analyzed (Participants) | 21
  Daily activities - change from week 8 to month 24 | 0.63 (14.206)
  Daily activities - from baseline to month 30: number analyzed (Participants) | 20
  Daily activities - from baseline to month 30 | 1.83 (18.621)
  Daily activities - from week 8 to month 30: number analyzed (Participants) | 20
  Daily activities - from week 8 to month 30 | 1.83 (15.652)
  Emotional impact - from baseline to month 24: number analyzed (Participants) | 21
  Emotional impact - from baseline to month 24 | 14.50 (19.130)
  Emotional impact - from week 8 to month 24: number analyzed (Participants) | 21
  Emotional impact - from week 8 to month 24 | 5.30 (13.905)
  Emotional impact - from baseline to month 30: number analyzed (Participants) | 20
  Emotional impact - from baseline to month 30 | 16.93 (19.710)
  Emotional impact - from week 8 to month 30: number analyzed (Participants) | 20
  Emotional impact - from week 8 to month 30 | 6.25 (15.761)
  Impact on work - from baseline to month 24: number analyzed (Participants) | 10
  Impact on work - from baseline to month 24 | 17.50 (37.657)
  Impact on work - from week 8 to month 24: number analyzed (Participants) | 9
  Impact on work - from week 8 to month 24 | -2.22 (16.976)
  Impact on work - from baseline to month 30: number analyzed (Participants) | 12
  Impact on work - from baseline to month 30 | 19.17 (29.835)
  Impact on work - from week 8 to month 30: number analyzed (Participants) | 11
  Impact on work - from week 8 to month 30 | -2.27 (11.481)
  Treatment effectiveness - from baseline to month 24: number analyzed (Participants) | 18
  Treatment effectiveness - from baseline to month 24 | 11.46 (27.390)
  Treatment effectiveness - from week 8 to month 24: number analyzed (Participants) | 18
  Treatment effectiveness - from week 8 to month 24 | 8.33 (20.895)
  Treatment effectiveness - from baseline to month 30: number analyzed (Participants) | 16
  Treatment effectiveness - from baseline to month 30 | 8.98 (27.192)
  Treatment effectiveness - from week 8 to month 30: number analyzed (Participants) | 17
  Treatment effectiveness - from week 8 to month 30 | 1.84 (28.791)
  Treatment bother/inconvenience - from baseline to month 24: number analyzed (Participants) | 20
  Treatment bother/inconvenience - from baseline to month 24 | -8.23 (24.756)
  Treatment bother/inconvenience - from week 8 to month 24: number analyzed (Participants) | 14
  Treatment bother/inconvenience - from week 8 to month 24 | -15.18 (28.241)
  Treatment bother/inconvenience - from baseline to month 30: number analyzed (Participants) | 19
  Treatment bother/inconvenience - from baseline to month 30 | 1.54 (19.243)
  Treatment bother/inconvenience - from week 8 to month 30: number analyzed (Participants) | 16
  Treatment bother/inconvenience - from week 8 to month 30 | -5.08 (21.677)
  Dry eye symptom-bother - from baseline to month 24: number analyzed (Participants) | 21
  Dry eye symptom-bother - from baseline to month 24 | -4.40 (15.571)
  Dry eye symptom-bother - from week 8 to month 24: number analyzed (Participants) | 21
  Dry eye symptom-bother - from week 8 to month 24 | -1.48 (18.143)
  Dry eye symptom-bother - from baseline to month 30: number analyzed (Participants) | 20
  Dry eye symptom-bother - from baseline to month 30 | -5.19 (14.579)
  Dry eye symptom-bother - from week 8 to month 30: number analyzed (Participants) | 20
  Dry eye symptom-bother - from week 8 to month 30 | -0.12 (11.691)

11. Secondary Outcome: Change From NGF0120 Baseline and NGF0120 Week 8 (EoT NGF0120=Baseline NGF0122) in Quality of Life Measured With EuroQol 5-Dimension 5-Level (EQ-5D-5L) to Months 24 and 30 of the NGF0122 Study.
Description: The EQ-5D-5L is a standardized questionnaire what measures the health status in 5 areas-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-with a rating scale of 1 (no problems) to 5 (extreme problems), where higher scores indicated worse problems.
  The questionnaire also asks the patient to rate their current health ("how good or bad your health is today") on a scale from 0 (worst health you can imagine) to 100 (best health you can imagine). On a 0-100 scale, a higher "your health today" score indicated better health. The EQ-5D-5L questionnaire was self-administered by the patient before any ophthalmic procedures at either visit.
  Please note that the severity level reported corresponds to the maximum experienced by the patient (for example, if a patient has one mild AE and one moderate AE, they are counted in the moderate category).
Time Frame: At Month 24 and Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
score on a scale
  Mobility - from Baseline to month 24: number analyzed (Participants) | 21
  Mobility - from Baseline to month 24 | -0.1 (0.62)
  Mobility - from week 8 to month 24: number analyzed (Participants) | 21
  Mobility - from week 8 to month 24 | -0.1 (0.54)
  Mobility - from Baseline to month 30: number analyzed (Participants) | 21
  Mobility - from Baseline to month 30 | 0.1 (0.94)
  Mobility - from week 8 to month 30: number analyzed (Participants) | 21
  Mobility - from week 8 to month 30 | 0.0 (0.59)
  Self-Care - from baseline to month 24: number analyzed (Participants) | 21
  Self-Care - from baseline to month 24 | 0.0 (0.32)
  Self-Care - from week 8 to month 24: number analyzed (Participants) | 21
  Self-Care - from week 8 to month 24 | -0.1 (0.54)
  Self-Care - from baseline to month 30: number analyzed (Participants) | 21
  Self-Care - from baseline to month 30 | 0.1 (0.65)
  Self-Care - from week 8 to month 30: number analyzed (Participants) | 21
  Self-Care - from week 8 to month 30 | 0.0 (0.67)
  Usual Activities - from baseline to month 24: number analyzed (Participants) | 21
  Usual Activities - from baseline to month 24 | -0.2 (0.83)
  Usual Activities - from week 8 to month 24: number analyzed (Participants) | 21
  Usual Activities - from week 8 to month 24 | 0.0 (0.55)
  Usual Activities - from baseline to month 30: number analyzed (Participants) | 21
  Usual Activities - from baseline to month 30 | -0.2 (0.93)
  Usual Activities - from week 8 to month 30: number analyzed (Participants) | 21
  Usual Activities - from week 8 to month 30 | 0.1 (0.83)
  Pain/Discomfort - from baseline to month 24: number analyzed (Participants) | 21
  Pain/Discomfort - from baseline to month 24 | -0.1 (0.77)
  Pain/Discomfort - from week 8 to month 24: number analyzed (Participants) | 21
  Pain/Discomfort - from week 8 to month 24 | -0.0 (0.67)
  Pain/Discomfort - from baseline to month 30: number analyzed (Participants) | 21
  Pain/Discomfort - from baseline to month 30 | -0.2 (0.87)
  Pain/Discomfort - from week 8 to month 30: number analyzed (Participants) | 21
  Pain/Discomfort - from week 8 to month 30 | -0.0 (0.86)
  Anxiety/Depression - from baseline to month 24: number analyzed (Participants) | 21
  Anxiety/Depression - from baseline to month 24 | -0.2 (1.14)
  Anxiety/Depression - from week 8 to month 24: number analyzed (Participants) | 21
  Anxiety/Depression - from week 8 to month 24 | -0.0 (1.02)
  Anxiety/Depression - from baseline to month 30: number analyzed (Participants) | 21
  Anxiety/Depression - from baseline to month 30 | -0.3 (0.86)
  Anxiety/Depression - from week 8 to month 30: number analyzed (Participants) | 21
  Anxiety/Depression - from week 8 to month 30 | -0.1 (0.83)

12. Secondary Outcome: Number/Percentage of Subjects Reporting Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the medicinal (investigational) product, whether or not related to the study product.
  AEs by severity (categorized as mild, moderate and severe) and relatedness (categorized as related and not related ) are considered - per each single subject - just once, at the greater severity and closest relationship to treatment. Considering that no study IMP was administered and that all standard of care were permitted, AEs must be read as related to any standard of care administered during the FU study.
Time Frame: From NGF0120 Week 8=NGF0122 Baseline to Month 30 of the NGF0122 study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Group Long-term Follow-up: All eligible patients in the original NGF0120 study, after completing enrollment, were invited to enter the Long-Term Follow-up Study (NGF0122) (all standard of care permitted), according to inclusion and exclusion criteria.
  The NGF0122 study aim was to assess the safety and efficacy of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophtalmic solution administered in Stage 1 Neurotrophic Keratitis patients enrolled in the original NGF0120 study. No intervention was performed in this extension study.
Arm/Group | Group Long-term Follow-up
Number analyzed (Participants) | 24
Participants
  number of patients reporting any AE | 20
  Number (%) of Subjects Reporting 0 AE | 4
  Number (%) of Subjects Reporting 1 AE | 2
  Number (%) of Subjects Reporting >1 AE | 18
  Number (%) of Subjects Reporting mild AEs | 5
  Number (%) of Subjects Reporting moderate AEs | 12
  Number (%) of Subjects Reporting severe AEs | 3
  Number (%) of Subjects Reporting AEs not related to any treatment administered | 14
  Number (%) of Subjects Reporting AEs related to any treatment administered | 6
  Number (%) of Subjects Reporting any serious AEs | 1

13. Secondary Outcome: Frequency of Normal and Clinically Significant Abnormal Findings for Slit-lamp Examination Parameters in the Study Eye at Baseline and Week 8 of the NGF0120 and at Month 24 and 30 of the NGF0122
Description: Slit-lamp biomicroscopy was performed in the study eye at Baseline and Week 8 of the NGF0120 study, and at Month 24 and 30. The anterior segment was evaluated under magnification using standard slit-lamp illumination. Parameters included eyelid edema and erythema, lashes, conjunctiva edema and bulbar erythema, cornea edema, endothelial and epithelial changes, lens, sclera, iris, and anterior chamber cells and flare. Findings were assessed visually as normal, abnormal not clinically significant, or abnormal clinically significant, based on clinical judgment and standard ophthalmologic criteria. Only the participants reporting normal and abnormal clinically significant results are shown (along with the percentage vs the "Number Analyzed", for each timepoint) The number of participants with abnormal not clinically significant results can be derived as difference between the sum of the said two categories and the "Number Analyzed", per each parameter and timepoint
Time Frame: Baseline and week 8 of the NGF0120, month 24 and 30 of the NGF0122
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group Long-term Follow-up - FAS
Number analyzed (Participants) | 24
Participants
  Lashes - Baseline - normal | 22
  Lashes - Baseline -abnormal CS | 0
  Lashes - week 8 - normal | 22
  Lashes - week 8 - abnormal CS | 0
  Lashes - month 24 - normal: number analyzed (Participants) | 21
  Lashes - month 24 - normal | 15
  Lashes - month 24 - abnormal CS: number analyzed (Participants) | 21
  Lashes - month 24 - abnormal CS | 3
  Lashes - month 30 - normal: number analyzed (Participants) | 21
  Lashes - month 30 - normal | 15
  Lashes - month 30 - abnormal CS: number analyzed (Participants) | 21
  Lashes - month 30 - abnormal CS | 3
  Eyelid Edema - Baseline - normal | 19
  Eyelid Edema - Baseline -abnormal CS | 0
  Eyelid Edema - week 8 - normal | 15
  Eyelid Edema - week 8 - abnormal CS | 0
  Eyelid Edema - month 24 - normal: number analyzed (Participants) | 21
  Eyelid Edema - month 24 - normal | 18
  Eyelid Edema - month 24 - abnormal CS: number analyzed (Participants) | 21
  Eyelid Edema - month 24 - abnormal CS | 1
  Eyelid Edema - month 30 - normal: number analyzed (Participants) | 21
  Eyelid Edema - month 30 - normal | 18
  Eyelid Edema - month 30 - abnormal CS: number analyzed (Participants) | 21
  Eyelid Edema - month 30 - abnormal CS | 3
  Eyelid Erythema - Baseline - normal | 20
  Eyelid Erythema - Baseline - abnormal CS | 1
  Eyelid Erythema - week 8 - normal | 19
  Eyelid Erythema - week 8 - abnormal CS | 1
  Eyelid Erythema - month 24 - normal: number analyzed (Participants) | 21
  Eyelid Erythema - month 24 - normal | 18
  Eyelid Erythema - month 24 - abnormal CS: number analyzed (Participants) | 21
  Eyelid Erythema - month 24 - abnormal CS | 1
  Eyelid Erythema - month 30 - normal: number analyzed (Participants) | 21
  Eyelid Erythema - month 30 - normal | 16
  Eyelid Erythema - month 30 - abnormal CS: number analyzed (Participants) | 21
  Eyelid Erythema - month 30 - abnormal CS | 1
  Conjunctiva Edema - Baseline - normal | 21
  Conjunctiva Edema - Baseline - abnormal CS | 0
  Conjunctiva Edema - week 8 - normal | 19
  Conjunctiva Edema - week 8 - abnormal CS | 1
  Conjunctiva Edema - month 24 - normal: number analyzed (Participants) | 21
  Conjunctiva Edema - month 24 - normal | 20
  Conjunctiva Edema - month 24 - abnormal CS: number analyzed (Participants) | 21
  Conjunctiva Edema - month 24 - abnormal CS | 0
  Conjunctiva Edema - month 30 - normal: number analyzed (Participants) | 21
  Conjunctiva Edema - month 30 - normal | 19
  Conjunctiva Edema - month 30 - abnormal CS: number analyzed (Participants) | 21
  Conjunctiva Edema - month 30 - abnormal CS | 0
  Conjunctiva Bulbar Erythema - Baseline - normal | 19
  Conjunctiva Bulbar Erythema - Baseline - abnormal CS | 0
  Conjunctiva Bulbar Erythema - week 8 - normal | 17
  Conjunctiva Bulbar Erythema - week 8 - abnormal CS | 2
  Conjunctiva Bulbar Erythema - month 24 - normal: number analyzed (Participants) | 21
  Conjunctiva Bulbar Erythema - month 24 - normal | 16
  Conjunctiva Bulbar Erythema - month 24 - abnormal CS: number analyzed (Participants) | 21
  Conjunctiva Bulbar Erythema - month 24 - abnormal CS | 1
  Conjunctiva Bulbar Erythema - month 30 - normal: number analyzed (Participants) | 21
  Conjunctiva Bulbar Erythema - month 30 - normal | 15
  Conjunctiva Bulbar Erythema - month 30 - abnormal CS: number analyzed (Participants) | 21
  Conjunctiva Bulbar Erythema - month 30 - abnormal CS | 2
  Corneal Epithelial Changes - Baseline - normal | 19
  Corneal Epithelial Changes - Baseline - abnormal CS | 2
  Corneal Epithelial Changes - week 8 - normal | 17
  Corneal Epithelial Changes - week 8 - abnormal CS | 4
  Corneal Epithelial Changes - month 24 - normal: number analyzed (Participants) | 21
  Corneal Epithelial Changes - month 24 - normal | 10
  Corneal Epithelial Changes - month 24 - abnormal CS: number analyzed (Participants) | 21
  Corneal Epithelial Changes - month 24 - abnormal CS | 5
  Corneal Epithelial Changes - month 30 - normal: number analyzed (Participants) | 21
  Corneal Epithelial Changes - month 30 - normal | 10
  Corneal Epithelial Changes - month 30 - abnormal CS: number analyzed (Participants) | 21
  Corneal Epithelial Changes - month 30 - abnormal CS | 5
  Corneal Endothelial Changes - Baseline - normal | 23
  Corneal Endothelial Changes - Baseline - abnormal CS | 0
  Corneal Endothelial Changes - week 8 - normal | 22
  Corneal Endothelial Changes - week 8 - abnormal CS | 1
  Corneal Endothelial Changes - month 24 - normal: number analyzed (Participants) | 21
  Corneal Endothelial Changes - month 24 - normal | 19
  Corneal Endothelial Changes - month 24 - abnormal CS: number analyzed (Participants) | 21
  Corneal Endothelial Changes - month 24 - abnormal CS | 2
  Corneal Endothelial Changes - month 30 - normal: number analyzed (Participants) | 21
  Corneal Endothelial Changes - month 30 - normal | 18
  Corneal Endothelial Changes - month 30 - abnormal CS: number analyzed (Participants) | 21
  Corneal Endothelial Changes - month 30 - abnormal CS | 2
  Cornea Edema - Baseline - normal | 24
  Cornea edema - Baseline - abnormal CS | 0
  Cornea Edema - week 8 - normal | 23
  Cornea Edema - week 8 - abnormal CS | 1
  Cornea Edema - month 24 - normal: number analyzed (Participants) | 21
  Cornea Edema - month 24 - normal | 20
  Cornea Edema - month 24 - abnormal CS: number analyzed (Participants) | 21
  Cornea Edema - month 24 - abnormal CS | 1
  Cornea edema - month 30 - normal: number analyzed (Participants) | 21
  Cornea edema - month 30 - normal | 21
  Cornea Edema - month 30 - abnormal CS: number analyzed (Participants) | 21
  Cornea Edema - month 30 - abnormal CS | 0
  Lens - Baseline - normal | 2
  Lens - Baseline - abnormal CS | 0
  Lens - week 8 - normal | 1
  Lens - week 8 - abnormal CS | 0
  Lens - month 24 - normal: number analyzed (Participants) | 21
  Lens - month 24 - normal | 1
  Lens - month 24 - abnormal CS: number analyzed (Participants) | 21
  Lens - month 24 - abnormal CS | 3
  Lens - month 30 - normal: number analyzed (Participants) | 21
  Lens - month 30 - normal | 2
  Lens - month 30 - abnormal CS: number analyzed (Participants) | 21
  Lens - month 30 - abnormal CS | 2
  Sclera - Baseline - normal | 24
  Sclera - Baseline - abnormal CS | 0
  Sclera - week 8 - normal | 24
  Sclera - week 8 - abnormal CS | 0
  Sclera - month 24 - normal: number analyzed (Participants) | 21
  Sclera - month 24 - normal | 21
  Sclera - month 24 - abnormal CS: number analyzed (Participants) | 21
  Sclera - month 24 - abnormal CS | 0
  Sclera - month 30 - normal: number analyzed (Participants) | 21
  Sclera - month 30 - normal | 21
  Sclera - month 30 - abnormal CS: number analyzed (Participants) | 21
  Sclera - month 30 - abnormal CS | 0
  Iris - Baseline - normal | 24
  Iris - Baseline - abnormal CS | 0
  Iris - week 8 - normal | 23
  Iris - week 8 - abnormal CS | 1
  Iris - month 24 - normal: number analyzed (Participants) | 21
  Iris - month 24 - normal | 20
  Iris - month 24 - abnormal CS: number analyzed (Participants) | 21
  Iris - month 24 - abnormal CS | 1
  Iris - month 30 - normal: number analyzed (Participants) | 21
  Iris - month 30 - normal | 19
  Iris - month 30 - abnormal CS: number analyzed (Participants) | 21
  Iris - month 30 - abnormal CS | 1
  Anterior Chamber Cells - Baseline - normal | 24
  Anterior Chamber Cells - Baseline - abnormal CS | 0
  Anterior Chamber Cells - week 8 - normal | 23
  Anterior Chamber Cells - week 8 - abnormal CS | 1
  Anterior Chamber Cells - month 24 - normal: number analyzed (Participants) | 21
  Anterior Chamber Cells - month 24 - normal | 20
  Anterior Chamber Cells - month 24 - abnormal CS: number analyzed (Participants) | 21
  Anterior Chamber Cells - month 24 - abnormal CS | 1
  Anterior Chamber Cells - month 30 - normal: number analyzed (Participants) | 21
  Anterior Chamber Cells - month 30 - normal | 21
  Anterior Chamber Cells - month 30 - abnormal CS: number analyzed (Participants) | 21
  Anterior Chamber Cells - month 30 - abnormal CS | 0
  Anterior Chamber Flare - Baseline - normal | 24
  Anterior Chamber Flare - Baseline - abnormal CS | 0
  Anterior Chamber Flare - week 8 - normal | 24
  Anterior Chamber Flare - week 8 - abnormal CS | 0
  Anterior Chamber Flare - month 24 - normal: number analyzed (Participants) | 21
  Anterior Chamber Flare - month 24 - normal | 21
  Anterior Chamber Flare - month 24 - abnormal CS: number analyzed (Participants) | 21
  Anterior Chamber Flare - month 24 - abnormal CS | 0
  Anterior Chamber Flare - month 30 - normal: number analyzed (Participants) | 21
  Anterior Chamber Flare - month 30 - normal | 21
  Anterior Chamber Flare - month 30 - abnormal CS: number analyzed (Participants) | 21
  Anterior Chamber Flare - month 30 - abnormal CS | 0

ADVERSE EVENTS:
Time Frame: For study participants enrolled in the NFG0120 study, the week 8 visit is the end of treatment visit and is to be considered as the baseline of the NGF0122 study. For the purpose of Adverse Events Reporting, the assessment period is from NGF0122 baseline (i.e., NGF0120 Week 8 / End of Treatment) till Month 30 of the NGF0122 study itself.
Groups:
- Group Long-term Follow-up - FAS: All eligible patients in the original NGF0120 study, after completing enrollment, were invited to enter the Long-Term Follow-up Study (NGF0122) (all standard of care permitted), according to inclusion and exclusion criteria.
  The NGF0122 study aim was to assess the safety and efficacy of OXERVATE® 0.002% (20 mcg/mL) cenegermin-bkbj ophtalmic solution administered in Stage 1 Neurotrophic Keratitis patients enrolled in the original NGF0120 study.
  No intervention was performed in this extension study.
Arm/Group | Group Long-term Follow-up - FAS
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Long-term Follow-up - FAS (N=24)
Pneumonia (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Long-term Follow-up - FAS (N=24)
Bradycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Corneal dystrophy (Congenital, familial and genetic disorders) | 3 (5)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 6 (12)
Eye pain (Eye disorders) | 4 (5)
Keratitis (Eye disorders) | 3 (5)
Vision blurred (Eye disorders) | 3 (4)
Eye irritation (Eye disorders) | 2 (4)
Neurotrophic keratopathy (Eye disorders) | 2 (4)
Blepharitis (Eye disorders) | 2 (3)
Cataract nuclear (Eye disorders) | 2 (3)
Punctate keratitis (Eye disorders) | 2 (3)
Corneal oedema (Eye disorders) | 1 (2)
Diplopia (Eye disorders) | 1 (2)
Eyelid irritation (Eye disorders) | 1 (2)
Ocular hypertension (Eye disorders) | 1 (2)
Ocular rosacea (Eye disorders) | 1 (2)
Open angle glaucoma (Eye disorders) | 1 (2)
Photopsia (Eye disorders) | 1 (2)
Presbyopia (Eye disorders) | 1 (2)
Vitreous adhesions (Eye disorders) | 1 (2)
Amblyopia (Eye disorders) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1)
Corneal deposits (Eye disorders) | 1 (1)
Corneal infiltrates (Eye disorders) | 1 (1)
Corneal scar (Eye disorders) | 1 (1)
Entropion (Eye disorders) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Trichiasis (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Secretion discharge (General disorders) | 1 (2)
Calcinosis (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Swelling face (General disorders) | 1 (1)
Graft versus host disease in lung (Immune system disorders) | 1 (1)
Graft versus host disease in skin (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Arthropod infestation (Infections and infestations) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (2)
Catheterisation cardiac (Investigations) | 1 (1)
Vital dye staining cornea present (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Overweight (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (3)
Migrane (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1)
Tonic clonic movements (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Tobacco user (Social circumstances) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1)
Transcatheter aortic valve implantation (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT05552261/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT05552261/SAP_001.pdf